CLINICAL TRIAL: NCT03171168
Title: The Effect of AposTherapy on Pain and Function in Knee Osteoarthritis Population: A Randomized Controlled Trial
Brief Title: The Effect of AposTherapy on Knee Pain
Acronym: AposKnee
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient recruitment and end of funding
Sponsor: Montefiore Medical Center (Other)
Collaborators: Apos Medical and Sports Technology Ltd. (Industry)
Responsible Party: Principal Investigator, Matthew Bartels, Professor and Chairman of Rehabilitation Medicine Albert Einstein College of Medicine, Montefiore Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015-4842
Record Dates: First submitted 2017-03-21; First posted 2017-05-31 (Actual); Results first posted 2022-12-14 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-11

CONDITIONS: Knee Osteoarthritis; Knee Pain
Keywords: Gait Analysis; WOMAC; SF-36 (Short Form 36)
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Single blinded (evaluator), single-center, randomized controlled trial. Interventional and Control group with option for Control group to Cross over.
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor is the only one masked in the study. Assessor is independent of the randomization, trial coordination, and care providers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Traditional Physical Therapy (Active Comparator): Participants will have traditional physical therapy up to 20 sessions, up to two sessions per week. This will involve exercise and modalities as decided by the therapists and medical providers. Participants will have a home exercise program for the remainder of the year.
  Interventions: Other: Traditional Physical Therapy
- AposTherapy (Experimental): Participants will have AposTherapy instead of traditional physical therapy over the course of one year. This will include 7 sessions of gait assessment and re-calibration with daily at home exercise with the device over the year.
  Interventions: Device: AposTherapy

INTERVENTIONS:
Device: AposTherapy — AposTherapy is a home-based exercise program utilizing footwear that causes exercise with normal daily activity that may significantly improve function in patients with knee pain in general, and specifically knee osteoarthritis (OA).
  Arms: AposTherapy
Other: Traditional Physical Therapy — Up to 20 sessions of traditional physical therapy
  Arms: Traditional Physical Therapy

SUMMARY:
AposTherapy is a home based exercise program utilizing footwear that causes exercise with normal activity that may significantly improve function in patients with knee osteoarthritis since patients with knee osteoarthritis have altered mechanics of motion contributing or due to the presence of the conditions. Capitalizing on the reported excellent adherence and clinical benefit of ApostTherapy in patients with significant knee OA, the investigators propose to evaluate this as a conservative treatment that may supplant/supplement traditional pain medications and physical therapy in an at-risk urban inner city population.

DETAILED DESCRIPTION:
AposTherapy is a home-based exercise program utilizing footwear that causes exercise with normal daily activity that may significantly improve function in patients with knee pain in general, and specifically knee osteoarthritis (OA). Capitalizing on the reported excellent adherence and clinical benefit of Apos Therapy in patients with significant lower limb arthritis, the investigators propose to evaluate this as a conservative treatment that may supplant/supplement traditional pain medications and physical therapy in knee OA population.

A potential use of AposTherapy as a replacement for traditional physical therapy may yield a less costly, more effective therapy with better adherence. Problems with traditional therapy include poor patient adherence (patients often do not complete the sessions and have very poor adherence (about 50-60%) to home therapy programs), added cost of travel (which may be more than $100 per session for ambulette or access-a-ride for eligible patients), and the lack of continuation in an ongoing exercise program, leading to relapse and need for retreatment. Additionally, access to physical therapy is limited for many patients since there are not enough available outpatient therapy services to meet the needs of all patients. Finding an alternative exercise program that will increase adherence, decrease total therapy visits, and improve patient's outcomes with decreased dependence on pain medications is a high priority from both patient care and cost management perspectives.

AposTherapy potentially overcomes many of these issues with improving/modifying abnormal biomechanics (therefore decreasing pain), and a home-based exercise program utilizing footwear that causes exercise with normal activity by promoting perturbation. This biomechanical approach may significantly reduce pain and improve function in patients with knee OA. Capitalizing on the reported excellent adherence and clinical benefit of AposTherapy in patients with significant knee OA, the investigators propose to evaluate the biomechanical exercise (wearing an appropriately calibrated shoe at home for a prescribed amount of time each day) as a conservative treatment that may supplement or supplant traditional pain medications, interventional pain procedures and physical therapy in an at-risk urban inner city population with knee OA.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from symptomatic knee OA (uni/bi lateral) for at least six months, fulfilling the American College of Rheumatology (ACR) clinical criteria for OA of the knee, and having radiographically assessed OA of the knee according to the Kellgren and Lawrence scale.
* Patients with a Visual Analog Scale (VAS) pain score of ≥3cm (measured at baseline).
* Males and females between the ages of 40-75.
* 17<BMI<40
* Ambulatory and active patients that can participate in a rehabilitation program that includes daily walking
* Stable medical regimen (no recent changes to the pain medication within a month)
* Able to walk at least 50 meters and scored positive on the STEADI test
* Able to understand, read and sign the informed consent form
* English or Spanish speaking

Exclusion Criteria:

* Patients suffering from acute septic arthritis.
* Patients suffering from inflammatory joint disease such as rheumatoid arthritis.
* Patients with diagnosis of avascular necrosis of the knee.
* Patients with diagnosis of neuromuscular disease.
* Patients with more than 3 falls in the last 12 months, OR any fall with an injury in the last 12 months.
* Patients exhibiting a lack of physical or mental ability to perform or comply with the study procedure.
* Patients with a history of pathological osteoporotic fracture
* Patients with referred pain in the knees from back or hip joint symptoms.
* Patients with severe back pain, ≥ 4 cm in visual analogue scale (0-10) [1] or radiating leg pain
* Patients with generalized body pain (both upper and lower extremities, such as fibromyalgia
* No major surgery to the affected limb and contralateral limb (e.g. no joint replacements or surgical fracture repair)
* No major cardiovascular comorbidities (able to enroll in an active exercise program)
* Patient started on lipid lowering medication in last 3 months
* Any change in blood pressure medications
* No recent physical therapy (no more recent than 6 months) on the affected limb
* No active heart disease (ischemia or heart failure admissions within 6 months) and no active Chronic Obstructive Pulmonary Disease (COPD) (exacerbation within 6 months)
* No active malignancies on ongoing treatment
* Patient with neurological gait pattern
* Patient requiring assistive device during gait analysis.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2016-11-30 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Bartels, MD, MPH, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center - Moses Campus, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jones KR, Vojir CP, Hutt E, Fink R. Determining mild, moderate, and severe pain equivalency across pain-intensity tools in nursing home residents. J Rehabil Res Dev. 2007;44(2):305-14. doi: 10.1682/jrrd.2006.05.0051. PMID 17551881
- [Background] Verghese J, Lipton RB, Hall CB, Kuslansky G, Katz MJ, Buschke H. Abnormality of gait as a predictor of non-Alzheimer's dementia. N Engl J Med. 2002 Nov 28;347(22):1761-8. doi: 10.1056/NEJMoa020441. PMID 12456852
- [Background] Elbaz A, Mor A, Segal G, Aloni Y, Teo YH, Teo YS, Das-De S, Yeo SJ. Patients with knee osteoarthritis demonstrate improved gait pattern and reduced pain following a non-invasive biomechanical therapy: a prospective multi-centre study on Singaporean population. J Orthop Surg Res. 2014 Jan 2;9:1. doi: 10.1186/1749-799X-9-1. PMID 24383821
- [Background] Haim A, Segal G, Elbaz A, Mor A, Agar G, Bar-Ziv Y, Beer Y, Morag G, Debi R, Atoun E. The outcome of a novel biomechanical therapy for patients suffering from anterior knee pain. Knee. 2013 Dec;20(6):595-9. doi: 10.1016/j.knee.2012.11.009. Epub 2012 Dec 27. PMID 23273535
- [Background] Drexler M, Elbaz A, Mor A, Debi R, Debbi EM, Haim A, Lador R, Salai M, Segal G. Effects of a customized biomechanical therapy on patients with medial compartment knee osteoarthritis. Ann Phys Rehabil Med. 2012 May;55(4):213-28. doi: 10.1016/j.rehab.2012.01.002. Epub 2012 Mar 27. English, French. PMID 22521468
- [Background] Segal G, Bar-Ziv Y, Velkes S, Benkovich V, Stanger G, Debbi EM, Debi R, Mor A, Elbaz A. A non-invasive biomechanical device and treatment for patients following total hip arthroplasty: results of a 6-month pilot investigation. J Orthop Surg Res. 2013 May 21;8:13. doi: 10.1186/1749-799X-8-13. PMID 23692690
- [Background] Forkan R, Pumper B, Smyth N, Wirkkala H, Ciol MA, Shumway-Cook A. Exercise adherence following physical therapy intervention in older adults with impaired balance. Phys Ther. 2006 Mar;86(3):401-10. PMID 16506876
- [Background] Sihvonen R, Paavola M, Malmivaara A, Itala A, Joukainen A, Nurmi H, Kalske J, Jarvinen TL; Finnish Degenerative Meniscal Lesion Study (FIDELITY) Group. Arthroscopic partial meniscectomy versus sham surgery for a degenerative meniscal tear. N Engl J Med. 2013 Dec 26;369(26):2515-24. doi: 10.1056/NEJMoa1305189. PMID 24369076
- [Background] Abbott JH, Robertson MC, Chapple C, Pinto D, Wright AA, Leon de la Barra S, Baxter GD, Theis JC, Campbell AJ; MOA Trial team. Manual therapy, exercise therapy, or both, in addition to usual care, for osteoarthritis of the hip or knee: a randomized controlled trial. 1: clinical effectiveness. Osteoarthritis Cartilage. 2013 Apr;21(4):525-34. doi: 10.1016/j.joca.2012.12.014. Epub 2013 Jan 8. PMID 23313532
- [Background] Fitzgerald GK, Hinman RS, Zeni J Jr, Risberg MA, Snyder-Mackler L, Bennell KL. OARSI Clinical Trials Recommendations: Design and conduct of clinical trials of rehabilitation interventions for osteoarthritis. Osteoarthritis Cartilage. 2015 May;23(5):803-14. doi: 10.1016/j.joca.2015.03.013. PMID 25952351
- [Background] Lim BW, Hinman RS, Wrigley TV, Sharma L, Bennell KL. Does knee malalignment mediate the effects of quadriceps strengthening on knee adduction moment, pain, and function in medial knee osteoarthritis? A randomized controlled trial. Arthritis Rheum. 2008 Jul 15;59(7):943-51. doi: 10.1002/art.23823. PMID 18576289
- [Background] Tanaka R, Ozawa J, Kito N, Moriyama H. Efficacy of strengthening or aerobic exercise on pain relief in people with knee osteoarthritis: a systematic review and meta-analysis of randomized controlled trials. Clin Rehabil. 2013 Dec;27(12):1059-71. doi: 10.1177/0269215513488898. Epub 2013 Jul 4. PMID 23828186
- [Background] Skou ST, Rasmussen S, Laursen MB, Rathleff MS, Arendt-Nielsen L, Simonsen O, Roos EM. The efficacy of 12 weeks non-surgical treatment for patients not eligible for total knee replacement: a randomized controlled trial with 1-year follow-up. Osteoarthritis Cartilage. 2015 Sep;23(9):1465-75. doi: 10.1016/j.joca.2015.04.021. Epub 2015 Apr 30. PMID 25937024

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Traditional Physical Therapy | AposTherapy
Started | 17 | 37
Completed | 10 | 19
Not Completed | 7 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Traditional Physical Therapy | AposTherapy | Total
Number analyzed (Participants) | 17 | 37 | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 23 | 36
  >=65 years | 4 | 14 | 18
Age, Continuous [Mean (Full Range); unit: years] | 59.24 [42 to 72] | 61.83 [47 to 78] | 61.01 [42 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 30 | 45
  Male | 2 | 7 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 16 | 25
  White | 0 | 5 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 7 | 15 | 22
Region of Enrollment [Number; unit: participants]
  United States | 17 | 37 | 54

OUTCOME MEASURES:

1. Primary Outcome: Knee Pain and Function
Description: Improvement in Pain and Function as assessed using the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) pain scale. The WOMAC, a self-administered instrument, is 1 of 3 subscales comprising the WOMAC Index. As a standalone measure, the WOMAC pain scale contains 5 items that address the following person-level activities: walking, using stairs, in bed, sitting or lying down, and standing upright. The stem of the scale asks the patient to focus on the extent of pain experienced in the involved knee during each of these activities which are reported on a 0-4 Likert scale: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4), with a possible score range of 0-20 for Pain. Higher scores on the WOMAC are associated with worse knee pain.
Time Frame: 24 weeks
Population: STUDY DISCONTINUED, statistical analysis was not performed due to study closure, not enough participants to conduct meaningful statistical analyses. The framework initially placed in the Statistical Analysis section has been removed. Analysis of individuals complete at 24 weeks. Only subjects with 24 week data were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Traditional Physical Therapy | AposTherapy
Number analyzed (Participants) | 8 | 30
units on a scale | 5.1 (2.8) | 3.2 (2.1)

2. Secondary Outcome: Quality of Life by RAND SF-36 (RAND Corporation Short Form 36)
Description: Health-related Quality of Life (QoL) as assessed using the RAND SF-36 (Short Form Health Survey). The RAND SF-36 is a 36-item patient-reported questionnaire that covers eight health domains: physical functioning (10 items), bodily pain (2 items), role limitations due to physical health problems (4 items), role limitations due to personal or emotional problems (4 items), emotional well-being (5 items), social functioning (2 items), energy/fatigue (4 items), and general health perceptions (5 items). Composite scoring range is 0 to 100 across the 8 domains identified with a higher overall score defining a more favorable health state.
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Traditional Physical Therapy | AposTherapy
Number analyzed (Participants) | 9 | 30
score on a scale | 48.8 (13.06) | 64.34 (16.0)

3. Secondary Outcome: PROMIS (Patient-Reported Outcomes Measurement Information System) Pain Interference and Physical Function
Description: Pain and Function measured through PROMIS short forms. PROMIS measures specific domains of Physical Health (e.g., physical function, pain intensity, pain interference, fatigue, sleep disturbance); Mental Health (depressive symptoms, anxiety, anger); and Social Health (ability to participate in social roles and activities).
  PROMIS measures are scored on the T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population. PROMIS domains use different terms to describe score ranges. For example, some domains use mild/moderate/severe whereas others use very high to very low. Cut points for assessment can also vary. For PROMIS measures, higher scores equals more of the concept being measured (e.g., more Fatigue, more Physical Function). Thus a score of 60 is one SD above the average referenced population. This could be a desirable or undesirable outcome.
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Traditional Physical Therapy | AposTherapy
Number analyzed (Participants) | 8 | 28
T-score | 20.7 (33.9) | 19.1 (41.9)

4. Secondary Outcome: Gait Assessment
Description: Objective assessment of the patients' gait assessed with gait analysis equipment. Equipment was used to measure the patients' cadence, or walking rate, in number of steps per minute (steps/min).
Time Frame: 24 weeks
Population: STUDY DISCONTINUED, statistical analysis was not performed due to study closure, not enough participants to conduct meaningful statistical analyses. Data presented is for patients who completed 24 weeks of the study. Data reported is only on those who entered the study and not outcomes data. Cadence is in steps per minute as entered below. As an example, typical marching is at 120 steps per minute.
Measure: Mean (Standard Deviation); unit: Cadence (steps/minute)
Arm/Group | Traditional Physical Therapy | AposTherapy
Number analyzed (Participants) | 12 | 27
Cadence (steps/minute) | 93.7 (20.1) | 109.7 (18.3)

5. Secondary Outcome: 6-min Walk Test
Description: objective assessment using maximum distance comfortably walked in 6 minutes on a 100 foot closed course
Time Frame: 24 weeks
Population: STUDY DISCONTINUED, statistical analysis was not performed due to study closure, not enough participants to conduct meaningful statistical analyses.
Measure: Mean (Standard Deviation); unit: Feet
Arm/Group | Traditional Physical Therapy | AposTherapy
Number analyzed (Participants) | 12 | 27
Feet | 1292 (229) | 1453 (228)

ADVERSE EVENTS:
Time Frame: 1 year
Description: No active intervention, only follow-up
Arm/Group | Traditional Physical Therapy | AposTherapy
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/37
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/37
Other Adverse Events (participants affected / at risk) | 5/17 | 10/37
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Traditional Physical Therapy (N=17) | AposTherapy (N=37)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Leg Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Back Pain (Nervous system disorders) | 0 (0) | 1 (1)
Inguinal hernia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Earache (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hyperkalemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Small Bowel Obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Umbilical hernia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cervical spondylosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lower Extemity Weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hypertension (Cardiac disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-26): https://cdn.clinicaltrials.gov/large-docs/68/NCT03171168/Prot_SAP_000.pdf